CLINICAL TRIAL: NCT00001446
Title: A Randomized Phase II Study of Oral Thalidomide in Patients With Hormone-Refractory Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 950178; 95-C-0178
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-08

CONDITIONS: Prostatic Neoplasm
Keywords: Angiogenesis; Malignancy; Neuropathy; Pharmacokinetics; Sedation
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Thalidomide

INTERVENTIONS:
Drug: thalidomide

SUMMARY:
This is a phase II study designed to evaluate the potential clinical efficacy of thalidomide in patients with hormone-refractory prostate cancer.

An important aspect of this study is to characterize the pharmacokinetics of thalidomide, as well as make correlations between the degree of angiogenesis occurring in a patient and the activity of thalidomide.

DETAILED DESCRIPTION:
This is a phase II study designed to evaluate the potential clinical efficacy of thalidomide in patients with hormone-refractory prostate cancer. Patients will be randomized to two different treatment arms (low dose versus high dose). An important aspect of this study is to characterize the pharmacokinetics of thalidomide, as well as make correlations between the degree of angiogenesis occurring in a patient and the activity of thalidomide. Each patient that has biopsiable lesions will undergo a pretreatment biopsy of their prostate (or other site of soft tissue disease) and repeat after 2 to 6 months of treatment. Additional information will be obtained on the changes in the circulating levels of the following growth factors: bFGF, TNF, VEGF, and TGFB. Neurological complications are the primary dose-limiting toxicity anticipated with chronic thalidomide administration.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Histologically documented adenocarcinoma of the prostate. Confirmation by the Clinical Center Pathology Department required.

CT-defined soft tissue disease required for staging if prostate-specific antigen (PSA) less than 20 ng/mL.

Progressive hormone-refractory disease for 1 month prior to entry (and after withdrawal of any antiandrogens), documented by at least one of the following: 3 consecutive rising levels of PSA at least 1 week apart. 1 measurement at least 50% greater than PSA nadir after last therapy.

New bone metastasis on Tc-99 bone scintigraphy.

Progression of measurable or evaluable soft-tissue metastases.

Development of new area of disease. 25% increase in previously measured lesions.

Total androgen ablation required. Testosterone in castrate range.

Concurrent luteinizing hormone-releasing hormone (LHRH) agonist required if not surgically castrated.

No prior prostate irradiation or radical prostatectomy unless other biopsiable lesions available.

Urgent local problems corrected prior to entry (e.g., severe bone pain, spinal cord compression, urinary flow obstruction).

No brain metastases.

PRIOR/CONCURRENT THERAPY:

Thyroid replaced concurrent to start of study for patients with chemical hypothyroidism.

Thyroid replaced prior to study for patients with clinical hypothyroidism.

Biologic Therapy: At least 4 weeks since Biologic Therapy and recovered from all toxic effects.

Chemotherapy:

No prior suramin.

At least 4 weeks since chemotherapy and recovered from all toxic effects.

Endocrine Therapy:

See Disease Characteristics.

At least 4 weeks since hormonal therapy except LHRH agonist therapy.

Radiotherapy:

See Disease Characteristics.

At least 4 weeks since radiotherapy (6 weeks since strontium).

Surgery: See Disease Characteristics.

PATIENT CHARACTERISTICS:

Age: 18 and over.

Performance status: ECOG 0-2.

Life expectancy: More than 3 months.

Hematopoietic:

Absolute granulocyte count greater than 1,000/mm(3).

Platelet count greater than 75,000/mm(3).

Hemoglobin greater than 8.0 g/dL (transfusion allowed if requirement maintained for more than 30 days OR bleeding identified and treated).

Hepatic:

Bilirubin no greater than 1.5 times normal.

AST and ALT less than 2.5 times normal.

Renal:

Creatinine no greater than 1.5 mg/dL OR

Creatinine clearance greater than 40 mL/min.

Proteinuria no greater than 2+ OR less than 500 mg/24 hr (except patients with ureteral stents).

BUN normal.

Electrolytes normal.

Urinalysis normal.

Cardiovascular:

No unstable or newly diagnosed angina.

No myocardial infarction within 6 months.

No NYHA class II-IV congestive heart failure.

Pulmonary:

No chronic obstructive lung disease requiring oxygen therapy.

Neurologic:

No clinically detectable peripheral neuropathy greater than grade 1.

No seizures within 10 years.

No anticonvulsants.

No requirement for sedatives or hypnotics.

OTHER:

Normal thyroid function tests at least 4 weeks prior to study and throughout study.

No concurrent anticoagulants.

No active infection.

Off antibiotics at least 1 week.

Ureteral stent or Foley catheter allowed with no antibiotics.

HIV negative.

No concurrent life-threatening illness.

No concurrent malignancies.

Ability to travel to the National Institutes of Health.

Adequate contraception required of sexually active patients and their partners during and for 2 months after therapy.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64
Dates: Start 1995-09; Study Completion 2001-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Bakay B, Nyhan WL. Binding of thalidomide by macromolecules in the fetal and maternal rat. J Pharmacol Exp Ther. 1968 Jun;161(2):348-60. No abstract available. PMID 5652850
- [Background] Barnhill RL, McDougall AC. Thalidomide: use and possible mode of action in reactional lepromatous leprosy and in various other conditions. J Am Acad Dermatol. 1982 Sep;7(3):317-23. doi: 10.1016/s0190-9622(82)70118-5. PMID 7130490
- [Derived] Sissung TM, Danesi R, Kirkland CT, Baum CE, Ockers SB, Stein EV, Venzon D, Price DK, Figg WD. Estrogen receptor alpha and aromatase polymorphisms affect risk, prognosis, and therapeutic outcome in men with castration-resistant prostate cancer treated with docetaxel-based therapy. J Clin Endocrinol Metab. 2011 Feb;96(2):E368-72. doi: 10.1210/jc.2010-2070. Epub 2010 Nov 24. PMID 21106711